CLINICAL TRIAL: NCT05581108
Title: Enhancement of Learning and Memory Following Supplementation With Juice PLUS+® OMEGA in an Adolescent Population
Acronym: AdCog-O
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Juice PLUS (Unknown)
Responsible Party: Principal Investigator, Prof Claire Williams, Professor, University of Reading
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RDG-007
Record Dates: First submitted 2022-06-13; First posted 2022-10-14 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Cognitive Change; Development, Adolescent
Keywords: Learning; Memory

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Juice PLUS+® OMEGA (Experimental): The Juice Plus+®Omega Blend capsules contain the following ingredients: DHA and EPAenriched oil of the micro algae Schizochytrium sp., pomegranate seed oil, coating agent: pullulan; raspberry seed oil, sea buckthorn oil 9, release agent: silicon dioxide; high oleic safflower seed oil, tomato seed oil, orange oil, vanilla oil, antioxidant: rosemary extract.
  Interventions: Dietary Supplement: Juice PLUS+® OMEGA
- Matched placebo (Placebo Comparator): Placebo capsules consist of medium chain triglycerides oil+ excipients like silicon dioxide aerosil, lecithin, vanilla flavor, orange oil, water and hypromellose(shell).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Juice PLUS+® OMEGA — Daily dose of total Omega blend: 925 mg (2 capsules)
  Arms: Juice PLUS+® OMEGA
Dietary Supplement: Placebo — matched placebo (2 capsules)
  Arms: Matched placebo

SUMMARY:
This study aims to investigate the effect of chronic supplementation with a commercially available, plant-derived, omega-3 intervention and cognitive performance in adolescent participants aged 13-14 years.

DETAILED DESCRIPTION:
A healthy diet is an essential factor for healthy ageing. Previous studies of omega-3 polyunsaturated fatty acids (n-3 PUFAs) intake have shown beneficial actions on a range of human health conditions. The influence of n-3 PUFAs on cognition throughout the lifespan is particularly apparent, with beneficial effects documented on cognitive development in infants and children, cognitive performance in young adults, and to slow age-related cognitive impairment in older adults. Despite these positive findings, there has been little consideration of the influence of n-3-PUFAs on cognition in adolescence. Adolescence is characterized by profound brain development, with brain areas such as the prefrontal cortex continuing to mature into the late twenties). In this period of brain development, the basis is laid for executive functions (e.g., shifting, updating, and short-term memory), among others. Optimal development of the prefrontal cortex is very important, as the executive functions have been related to academic achievements. The positive effects from n-3 PUFAs on cognition, if translated to adolescents, would be of clear practical and theoretical importance, particularly in an academic context.

￼

This project will examine the relationship between supplementation with a commercially available, plant-derived, omega-3 intervention and cognitive performance in adolescent participants aged 13-14 years. In a randomized, placebo-controlled, double-blind, parallel-group clinical trial, we will examine the effect of 16 weeks repeated daily dosing of Juice PLUS+® OMEGA (or matched placebo) on a wide range of cognitive processes (measured using a battery of computer-based cognitive tests). Changes in cognitive performance will be mapped both to changes in omega-3 index (O3I) of our participants (measured using dried blood spots obtained via finger prick) and to changes in brain activity (measured using electrodes placed on the scalp, in a subset of participants). Participants will attend the Department on 3 separate occasions. At an initial screening visit, participants will practice the cognitive tests and provide a 3-day food diary as a measure of habitual diet. Participants will then attend a baseline test visit, where they will perform the cognitive tests and receive a 16-week supply of capsules (either placebo or active treatment) to be taken daily. After the 16 weeks, the participants will attend a post-intervention test day where they will perform the cognitive tests for a final time. Finger prick blood spot samples will be taken at each of the 3 visits.

ELIGIBILITY:
Inclusion Criteria:

* age 13-14, fruit and vegetable intake less than or equal to 3 servings per day, not more than 2 servings of fish per week, English as a first language, adequate visual and auditory acuity to perform the cognitive tasks, normal BMI for age, normal British Ability Scales (BAS) score

Exclusion Criteria:

* psychological or psychiatric disorders, ADHD or dyslexia diagnosis, fruit/vegetable or histamine intolerance, use of medications or dietary supplements that may impact study outcomes, conditions altering absorption of nutrients (e.g. celiac disease), antibiotic use within the last 3 months, adherence to any specific diets that may impact study outcomes (e.g. vegetarian, paleo etc.

Ages: 13 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
Rate of Learning (Rey Auditory Verbal Learning Task) | Baseline
  Participants will be presented with a sequential list of 15 words, at a rate of 1 word per second. The participant will then have 60s to say out loud as many of these words as possible, with the resulting score recorded as a percentage of accuracy. This occurs 5 times for the same word list, and the rate of learning is determined through change in accuracy across the 5 recalls.
Rate of Learning (Rey Auditory Verbal Learning Task) | 16 weeks
  Participants will be presented with a sequential list of 15 words, at a rate of 1 word per second. The participant will then have 60s to say out loud as many of these words as possible, with the resulting score recorded as a percentage of accuracy. This occurs 5 times for the same word list, and the rate of learning is determined through change in accuracy across the 5 recalls.
Delayed Word Recall (Rey Auditory Verbal Learning Task) | Baseline
  After a period of time subject are asked to recall as many words as possible from list A
Delayed Word Recall (Rey Auditory Verbal Learning Task) | 16 weeks
  After a period of time subject are asked to recall as many words as possible from list A
Word Recognition (Rey Auditory Verbal Learning Task) | Baseline
  Following the delayed word recall, words from list A, list B and novel words are displayed sequentially on the screen and participants are asked to indicate which words were from list A only.
Word Recognition (Rey Auditory Verbal Learning Task) | 16 weeks
  Following the delayed word recall, words from list A, list B and novel words are displayed sequentially on the screen and participants are asked to indicate which words were from list A only.

SECONDARY OUTCOMES:
Change in Modified Attention Network Task (MANT) | 16 weeks
  This task examines execution function, attention and inhibition. In this task, participants have to respond to a centrally presented arrow, pointing to the left or the right by pressing the corresponding key on the keyboard. The central arrow is flanked by arrows that point in the same (congruent) or opposite (incongruent) direction. In order to perform the task effectively, participants have to ignore the flanking arrows. Previous studies have found that participants show larger latencies and more errors on incongruent trials when compared with congruent trials due to the conflicting interference of the incongruently facing arrows. The response latencies to congruent trials reflect processing speed, while the amount of interference during incongruent trials indicates susceptibility to interference.
Change in N-Back | 16 weeks
  The N-Back task is a measure of working memory where participants are instructed to monitor a series of stimuli and to respond whenever a stimulus is presented that is the same as the one presented n trials previously. In this simplified 0-back version, participants respond when the target matches a fixed target specified at the beginning of the task (similar to a Go/No-Go task). Data will be analysed for both accuracy and reaction time on correct trials. For a subset of participants, this task will be conducted while recording EEG in order to monitor change in brain activity in response to target trials. The N-Back was selected as it has been shown in previous work to elicit a strong P300 signal (see EEG as additional outcome).
Change in PANAS-c | 16 weeks
  A validated self-report measure of affective state in children. The PANAS comprises of two distinct affective states (positive and negative), as well as 11 individual affective states (fear, guilt, sadness, surprise, hostility, shyness, joviality, self-assurance, attentiveness, fatigue and serenity. Subjects use a likert scale from 1 - 5 to indicate how the word relates to how they are currently feeling.
Change in Task Switching Test (TST) | 16 weeks
  This task requires executive function and sustained attention, and provides a measure of cognitive flexibility. Participants view a circle with 8 equally spaced radii 2 of which form a bold bisecting line. Numbers are chosen randomly from a set of 1-4 & 6-9 and displayed sequentially in a clockwise direction. A response of higher or lower than 5 is made for trials below the bold line, and even or odd for numbers above the line. Outcome measures include overall accuracy and reaction time (RT) on correct trials, as well as accuracy and RT on trials where there is a 'switch cost' from stimuli moving from below to above the bold line and vice versa.
Change in Emotion Regulation Questionnaire for Children and Adults (ERQ-CA) | 16 weeks
  A validated 10-item questionnaire used to assess emotion regulation, specifically reappraisal and suppression.

OTHER OUTCOMES:
Change in P300 | 16 weeks
  Change in ERP measure of P300 latency and amplitude will be assessed using EEG (electroencephalography) in a subset of participants during resting state (eyes open and closed) and during the N-Back task. EEG data will be collected using Brain Products software and 16-channel active electrodes.
Change in Omega 3 Index | 16 weeks
  Finger-prick dried blood spots will be collected before and after omega 3 supplementation to assess change in fatty acid profile in red blood cell membranes. Analysis will be performed by Omega Quant.
Change in Power Spectral Density (PSD) | 16 weeks
  Changes in Power for Alpha, Beta, Gamma, Delta, and Theta bands during performance of the N-Back task.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Williams, Prof, Principal Investigator — University of Reading
Locations (1):
- School of Psychology and Clinical Languages, University of Reading, Reading, Berkshire, United Kingdom

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-08-15): https://cdn.clinicaltrials.gov/large-docs/08/NCT05581108/SAP_000.pdf